CLINICAL TRIAL: NCT04579965
Title: Misotac vs Combined Oral Contraceptive Pill in the Treatment of Symptomatic Isthmocele
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Alaa Wageh, Alaa Wageh Associate Professor Obstetrics and gynecology, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Dysfunctional Uterine Bleeding
Keywords: Postmenstrual bleeding; Isthmocele; Combined Oral Contraceptive Pill; Misotac
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined contraceptive pills (Other): treat patients with isthmocele with oral contraceptive pills
  Interventions: Drug: medical treatment of isthmocele
- Misotac (Other): treat patients with isthmocele with misotac.
  Interventions: Drug: medical treatment of isthmocele

INTERVENTIONS:
Drug: medical treatment of isthmocele — comparison between different drugs

SUMMARY:
Isthmocele is a growing concern as a cause of abnormal uterine bleeding, especially post menstrual bleeding which may be present in up to 82% of these cases (Iannone et al 2019).

our trial is a randomized clinical trial in which women will be randomly allocated to either medical treatment by oral contraceptive or to medical treatment by misotac.

DETAILED DESCRIPTION:
Isthmocele is a growing concern as a cause of abnormal uterine bleeding, especially post menstrual bleeding which may be present in up to 82% of these cases There is no universal standard definition of isthmocele but most of the authors agree that isthmocele as a myometrial discontinuity in the myometrium of the anterior uterine wall of >2mm at the site of a cesarean scar in non-pregnant women.

Treatment should be offered only to the symptomatic patient. Surgery, by hysteroscopy, laparoscopy, laparotomy, or vaginal routes, is the most common treatment of choice even in the small defect Surgery is not without complications and many women reject it as a treatment option so it is reasonable to look for medical methods of management.

The pathogenesis of AUB following the development of isthmocele remains unexplained. Oral contraceptive pills might represent a valid option due to a regulatory effect on the endometrium. Several authors describe the effectiveness of oral contraceptives in reducing bleeding disorders correlated to isthmocele.

Another theory of AUB following the development of isthmocele is that menstrual blood can be collected in the defect so that it seeps slowly over the days following menstruation. This mechanism is added by impaired uterine contractility at the scar area.

Misoprostol is a synthetic analog of prostaglandin E1, which increases myometrial contractions so it can be used for various other indications in obstetrics and gynecology the aim is to examine two different methods of medical treatment in cases of symptomatic isthmocele; first regulatory effect on the endometrium (Oral contraceptive pills) and second contraction of myometrium (misotac)

Patient and methods:

Women with a previous cesarean section who presented with postmenstrual spotting, and in whom sonohysterography had shown a isthmocele were eligible. A isthmocele was defined as an indentation in the anterior uterine wall at the site of the caesarean scar with at least 2 mm depth, measured during sonohysterography.

Postmenstrual spotting needed to be present for at least three consecutive months after the last cesarean section. Postmenstrual spotting was defined as two or more days of brownish discharge at the end of menstrual bleeding when the total period of menstrual bleeding exceeds 7 days

Exclusion criteria included any organic condition that will be the cause of that bleeding; Pregnancy, (suspected) malignancies, use of any hormonal contraceptives, fibroid, infection in the genital tract, etc.

Randomization After written informed consent was given, women were randomly allocated to either medical treatment by oral contraceptive or to medical treatment by misotac.

ELIGIBILITY:
Inclusion Criteria:

* Women with a previous cesarean section
* who presented with postmenstrual spotting,
* sonohysterography had shown a isthmocele

Exclusion Criteria:

* Pregnancy,
* (suspected) malignancies,
* use of any hormonal contraceptives,
* fibroid,
* infection in the genital tract

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
postmenstrual spotting. | after one month of drug treatment
  the effect of the drugs on the number of days with postmenstrual spotting during a menstrual cycle.

SECONDARY OUTCOMES:
Quality of life, Satisfaction assessed by the VAS | after one month of drug treatment
  the effect of the drugs on Quality of life, Satisfaction

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iannone P, Nencini G, Bonaccorsi G, Martinello R, Pontrelli G, Scioscia M, Nappi L, Greco P, Scutiero G. Isthmocele: From Risk Factors to Management. Rev Bras Ginecol Obstet. 2019 Jan;41(1):44-52. doi: 10.1055/s-0038-1676109. Epub 2019 Jan 15. PMID 30646424
- [Background] Kremer TG, Ghiorzi IB, Dibi RP. Isthmocele: an overview of diagnosis and treatment. Rev Assoc Med Bras (1992). 2019 Jun 3;65(5):714-721. doi: 10.1590/1806-9282.65.5.714. PMID 31166450
- [Background] Zhang X, Yang M, Wang Q, Chen J, Ding J, Hua K. Prospective evaluation of five methods used to treat cesarean scar defects. Int J Gynaecol Obstet. 2016 Sep;134(3):336-9. doi: 10.1016/j.ijgo.2016.04.011. Epub 2016 Jun 30. PMID 27473332
- [Background] Florio P, Gubbini G, Marra E, Dores D, Nascetti D, Bruni L, Battista R, Moncini I, Filippeschi M, Petraglia F. A retrospective case-control study comparing hysteroscopic resection versus hormonal modulation in treating menstrual disorders due to isthmocele. Gynecol Endocrinol. 2011 Jun;27(6):434-8. doi: 10.3109/09513590.2010.495431. Epub 2011 Jan 4. PMID 21204608
- [Background] Tahara M, Shimizu T, Shimoura H. Preliminary report of treatment with oral contraceptive pills for intermenstrual vaginal bleeding secondary to a cesarean section scar. Fertil Steril. 2006 Aug;86(2):477-9. doi: 10.1016/j.fertnstert.2006.01.020. Epub 2006 Jun 12. PMID 16769058
- [Background] Thurmond AS, Harvey WJ, Smith SA. Cesarean section scar as a cause of abnormal vaginal bleeding: diagnosis by sonohysterography. J Ultrasound Med. 1999 Jan;18(1):13-6; quiz 17-8. doi: 10.7863/jum.1999.18.1.13. PMID 9952074
- [Background] Wu HL, Marwah S, Wang P, Wang QM, Chen XW. Misoprostol for medical treatment of missed abortion: a systematic review and network meta-analysis. Sci Rep. 2017 May 10;7(1):1664. doi: 10.1038/s41598-017-01892-0. PMID 28490770
- [Background] Tower AM, Frishman GN. Cesarean scar defects: an underrecognized cause of abnormal uterine bleeding and other gynecologic complications. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):562-72. doi: 10.1016/j.jmig.2013.03.008. Epub 2013 May 14. PMID 23680518
- [Background] Vervoort A, van der Voet LF, Hehenkamp W, Thurkow AL, van Kesteren P, Quartero H, Kuchenbecker W, Bongers M, Geomini P, de Vleeschouwer L, van Hooff M, van Vliet H, Veersema S, Renes WB, Oude Rengerink K, Zwolsman SE, Brolmann H, Mol B, Huirne J. Hysteroscopic resection of a uterine caesarean scar defect (niche) in women with postmenstrual spotting: a randomised controlled trial. BJOG. 2018 Feb;125(3):326-334. doi: 10.1111/1471-0528.14733. Epub 2017 Jul 5. PMID 28504857